CLINICAL TRIAL: NCT05537584
Title: SMART Trial to Predict Anhedonia Response to Antidepressant Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Diego Pizzagalli, Professor, Department of Psychiatry, Harvard Medical School, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022P000896
Record Dates: First submitted 2022-09-06; First posted 2022-09-13 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sertraline; Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MDD with SERT+ Response Marker (Experimental): Participants with MDD who have been classified as high sertraline responders based on behavioral and brain data.
  Interventions: Drug: Sertraline; Drug: Bupropion
- MDD with BUP+ Response Marker (Experimental): Participants with MDD who have been classified as high bupropion responders based on behavioral and brain data.
  Interventions: Drug: Sertraline; Drug: Bupropion

INTERVENTIONS:
Drug: Sertraline — Subjects will receive 8 weeks of sertraline while monitored by the study physician
  Other Names: Zoloft
Drug: Bupropion — Subjects will receive 8 weeks of bupropion while monitored by the study physician
  Other Names: Wellbutrin

SUMMARY:
The main goal of this research is to use behavioral, brain, and clinical data to determine which type of antidepressant might be optimal before people with depression start treatment.

DETAILED DESCRIPTION:
The treatment of depression is often trial-and-error. Earlier research reported that only 50% of individuals with depression show a significant decline in symptoms after taking an antidepressant. The situation is even worse in primary care, where only 30% respond to first line antidepressants.

The difficulty in treating depression is likely because treatment selection is not based on each person's characteristics. While some depressed individuals may benefit from selective serotonin reuptake inhibitors (SSRIs), others might benefit more from other types of medication. Finding markers that predict an individual's response to different antidepressants would provide patients and clinicians with valuable information to guide treatment selection.

The present study is among the first to use clinical (e.g., responses on questionnaires), behavioral (e.g., performance in computerized tasks), and brain (e.g., MRI scans) data to guide treatment selection in order to increase the likelihood of benefiting from one of two antidepressants. After analyzing an individuals' markers, subjects will be randomly assigned to receive a full 8-week course of an SSRI or non-SSRI.

Throughout the study, participants will complete 9 total sessions over the course of 9-10 weeks, including an electroencephalogram (EEG) recording, a functional magnetic resonance imaging (fMRI) scan, an electrocardiogram (EKG) exam, interviews with clinicians, and a full 8-week course of an antidepressant.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 64
* Any gender and all ethnic/racial origins
* Diagnosis of Major Depressive Disorder. MDD diagnosis will be decided by clinicians via the Structured Clinical Interview for DSM-5 (SCID-5).
* Elevated depression severity
* Elevated anhedonia symptoms
* Fluency in written and spoken English
* Ability to give signed, informed consent either written or electronic
* Normal or corrected-to-normal vision and hearing
* Ability to adhere to the study schedule

Exclusion Criteria:

* Patient is currently enrolled in any treatment program except psychotherapy (transcranial magnetic stimulation, other antidepressants etc.).
* Any contraindication to bupropion or sertraline considered unsafe by the study physician, or any history of adverse reaction to either drug.
* Failure to respond to an adequate course of treatment with both of the study medications (sertraline or bupropion) during the current episode.
* Participants who are determined to be treatment resistant, (i.e., having failed to respond to at least two adequate antidepressant trials in the current episode)
* Pregnant women, or women of childbearing potential who have a positive result on a urine pregnancy test
* Failure to meet MRI safety requirements, including any metal implants or prostheses that cannot be removed, or exposure to shrapnel
* Claustrophobia or severe anxiety that might affect participation in neuroimaging
* Injury or movement disorder that may make it difficult to lie still in the scanner
* Any current recreational/illicit drug use, with the exception of THC, as assessed by a urine drug test (covering cocaine, cannabinoids, opiates, amphetamines, methamphetamines, phencyclidine, MDMA, benzodiazepines, methadone, oxycodone, tricyclic antidepressants, and barbiturates). Participants who use THC regularly will be allowed to continue in the study provided they have abstained for the three days prior to visits involving the MRI scan.
* Use of Monoamine Oxidase Inhibitors (MAOIs) either currently or within the past two weeks
* Participants who are currently stopping the use of tobacco products. Participants who cannot abstain from tobacco products for eight hours without cravings.
* More than 15 alcohol-induced lifetime blackouts.
* History of regular use (5-7xs per week) of marijuana before the age of 15
* Lifetime history of other recreational drug use beyond the following limits (for each drug individually) and/or last use within the past 3 months:

  1. Hallucinogens (mushrooms, LSD): exclude for12 uses in the past year, or 15 uses lifetime (unless last use was 5+ years ago, then allow up to 25 lifetime uses)
  2. Ecstasy: exclude for 12 uses in the past year, or 15 uses lifetime (unless last use was 5+ years ago, then allow up to 25 lifetime uses)
  3. Anxiolytics (recreational use): exclude for 12 uses in the past year, or 15 uses life time (unless last use was 5+ years ago, then allow up to 25 lifetime uses)
  4. Cocaine, meth/psychostimulants (this includes prescribed stimulants such as methylphenidate) exclude for 5 uses in the past year, or 10 uses lifetime
  5. Prescribed opioids for a limited period (e.g., post-surgery) is OK if no use in the past 3 months
  6. 3 uses: Inhalants, IV drugs, crack cocaine, or crystal methamphetamine
* Recent use (within 3 weeks) of any medication that affects blood flow or blood pressure, or which is vasodilating/vasoconstricting (for participants undergoing neuroimaging)
* Metformin use in the past 6 months (for either clinical care or as part of research)
* Serious or unstable medical illness
* Current infectious illness (either transient or chronic); Current episode of allergic reaction or asthma
* Hemophilia; Diabetes with poor glucose control; History of chronic migraine (> 15 days/mo.); History of dementia.
* History of seizures or seizure disorder.
* Any history of significant head injury or concussion with loss of consciousness for two minutes or more, or head injury with lingering functional/psychological impact
* Serious structural cardiac abnormalities, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems (contraindication to bupropion)- confirmed with ECG at physicians' discretion.
* Past/current DSM-5 diagnosis of: OCD, schizophrenia or other psychotic disorders, schizoaffective disorder, delusional disorder, psychotic disorders NOS, bipolar disorder, patients with mood congruent or mood incongruent psychotic features, autism or any other pervasive developmental disorder, organic mental disorder, PTSD (current only), somatoform disorder, severe borderline or antisocial personality disorder, anorexia or current subthreshold anorexia, binge eating disorder, or bulimia (however bulimia is allowed if it has been fully remitted in the past 2 years; binge eating disorder is allowable if it has been partially remitted within the past 3 months; current subthreshold binge eating disorder is allowable; past PTSD fully remitted for longer than one month and current partial remission of PTSD is allowable)
* Current mild, moderate, or severe substance (including cannabis) or alcohol use disorder. Early or sustained remission is allowable, i.e., criteria for any level of abuse has not been met for at least the past 3 months (with the exception of past or current cocaine, stimulant, or opioid abuse, which will lead to automatic exclusion).
* Specific phobia, social anxiety disorder and generalized anxiety disorders will be allowed only if judged to be currently mild and never the principal diagnosis when co-occurring with current or past MDD. Panic disorder will be allowed if MDD is the principal diagnosis and panic disorder has been in remission for > 2 years.
* Electroconvulsive Therapy in the current episode.
* Patient is clinically unstable, in the judgment of the clinician or physician.
* Participants with suicidal ideation where continued study participation is believed unsafe by the study clinician or study physician (these participants will be immediately referred to appropriate clinical treatment).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Score on Montgomery-Asberg Depression Rating Scale (MADRS) | 8-10 weeks
  Symptoms of depression

SECONDARY OUTCOMES:
Ventral-striatal activation during reward related tasks in an fMRI scan | 8-10 weeks
  Brain measure of anhedonia
Effort-based decision making during an effort-based task | 8-10 weeks
  Behavioral measure of anhedonia
Reward positivity during a guessing monetary reward task | 8-10 weeks
  Behavioral measure of anhedonia
Cortico-insular activation during an effort-based task | 8-10 weeks
  Brain measure of anhedonia
Resting state functional connectivity between the NAc and mPFC during an fMRI scan | 8-10 weeks
  Brain measure of anhedonia

CONTACTS AND LOCATIONS:
Overall Officials: Diego A. Pizzagalli, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
We are part of a large team of researchers across the US called MCPsych which is funded through the Wellcome Leap Grant. We have a large repository of questionnaires, behavioral, and brain data that will be collected similar across sites and allow additional data analyses.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 12 months after data collection is completed
Access Criteria: Access will be governed by the Multi-Channel Psych department of the Wellcome Leap foundation.